CLINICAL TRIAL: NCT02838888
Title: Computer-assisted Detection of Colonic Polyps
Acronym: KoloPol I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Fraunhofer Institut Erlangen (Unknown)
Responsible Party: Sponsor
Other Study IDs: KoloPol I
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Colon Adenoma
Keywords: Adenoma; computer; automatic; polyp; detection
MeSH Terms: conditions — Adenoma; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colon polyps
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Routine colonoscopy Cohort: Patients receiving routine colonoscopy at the study site
  Interventions: Device: Automatic polyp detection software

INTERVENTIONS:
Device: Automatic polyp detection software — A computer program for the detection of colonic polyps will be used during colonoscopy

SUMMARY:
Screening colonoscopy is considered the gold standard for adenoma detection in the colon. However, it has been shown that a considerable number of polyps can be missed during screening colonoscopy. Until now the endoscopist himself is responsible for the detection of adenomatous polyps. No automatic tools are available supporting the colonoscopist to detect lesions. Recently, a computer program was developed that can be used to recognize and extract suspicious structure from colonoscopy video sequences. The program was built to automatically detected colonic polyps and to highlight the polyps by colour marking. The program was now refined so that the respective structures can be highlighted during real time colonoscopy. The aim of this feasibility study is to test whether the software is applicable during real time colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Indication for colonoscopy
* age ≥ 40 years

Exclusion Criteria:

* American Society of Anesthesiologists class IV or higher
* pregnant women
* indication for colonoscopy: inflammatory bowel disease
* indication for colonoscopy: polyposis syndrome
* indication for colonoscopy: emergency colonoscopy e.g. acute bleeding

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving colonoscopy at the study site are eligible for participation.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Polyp detection | up to 2 weeks (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks)
  After obtaining the histopathological diagnosis of resected polyps (approximately 3 days - 2 weeks) it can be determined whether the resected specimen contained polyp histology or not.

CONTACTS AND LOCATIONS:
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klare P, Sander C, Prinzen M, Haller B, Nowack S, Abdelhafez M, Poszler A, Brown H, Wilhelm D, Schmid RM, von Delius S, Wittenberg T. Automated polyp detection in the colorectum: a prospective study (with videos). Gastrointest Endosc. 2019 Mar;89(3):576-582.e1. doi: 10.1016/j.gie.2018.09.042. Epub 2018 Oct 17. PMID 30342029